CLINICAL TRIAL: NCT02037009
Title: Centralised Anesthesic Monitoring in the Surgery of the Ocular Anterior Segment: Non Inferiority Study
Acronym: SACHS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fondation Ophtalmologique Adolphe de Rothschild (Network)
Collaborators: Ministry of Health, France (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: SC_JMD_2013-1
Record Dates: First submitted 2014-01-13; First posted 2014-01-15 (Estimated); Last update posted 2026-01-06 (Actual); Status verified 2026-01

CONDITIONS: Ambulatory Surgical Procedures; Ocular Anterior Segment Surgery

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Usual surveillance (No Intervention): surveillance performed by a qualified nurse, present in the operating room during the whole anesthesia.
- centralised monitoring surveillance (Experimental): 1 anesthetic nurse is posted at a centralised monitoring station outside of the 3 operating rooms, while another one can intervene inside the 3 operating rooms whenever needed. Interphones allow communication between the monitoring station and the operating rooms.
  Interventions: Other: Health care organization (anesthetic surveillance)

INTERVENTIONS:
Other: Health care organization (anesthetic surveillance)
  Arms: centralised monitoring surveillance

SUMMARY:
In France, cataract surgery is the most frequent surgical procedure, performed with local anesthesia and most often very light techniques using eye-drops. Technical improvements of surgical and anesthesic procedures have led many countries to implement alternative surveillance procedures. In France, it is mandatory that the persons in charge of anesthetic surveillance (doctors or nurses) should be qualified in anesthesia.

In this study, the investigators aim to assess the feasibility and safety of a centralised monitoring station outside of the operating rooms, as an alternative to the presence of 1 anesthetic nurse in each operating room.

DETAILED DESCRIPTION:
In their hospital, the investigators will study the following alternatives for the anesthetic surveillance of the 3 operating rooms where surgery of the ocular anterior segment is performed: 1) the usual procedure, with the presence of 3 anesthetic nurses (1 in each operating room) and 2) a new organization with an anesthetic nurse checking a centralised monitoring station and a back-up anesthetic nurse ready to intervene inside the 3 operating rooms whenever needed.

The 2 procedures will be successively implemented during 3 to 4 sequences, until the number of surgical procedures statistically required have been studied.

The investigators aim to demonstrate that the centralised monitored surveillance does not put the patients at risk more often than the current surveillance procedure.

ELIGIBILITY:
Inclusion Criteria:

* adult patient scheduled for ocular anterior segment surgery (cataract, glaucoma, pterygium) with local or topic anesthesia

Exclusion Criteria:

* patient refusing to participate in the study or without health insurance

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 900 (Actual)
Dates: Start 2013-11; Primary Completion 2014-04 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Anesthetic potential impact on surgery conditions | during surgical procedure
  Incidence rate of at least 1 of the following events, during surgery:
  * blood pressure > 200 mmHg on 2 consecutive measures (automatic measure every 3 minutes)
  * cardiac frequency < 45/min for at least 1 mn
  * SaO2 <85% for at least 1 mn
  * poor operating conditions (rated ≤ 7 by the surgeon, on a numeric scale from 0 to 10=excellent conditions). Assessment at the exit of operating room.

SECONDARY OUTCOMES:
interventions of the back-up anesthetic nurse | during surgical procedure
  mean number of interventions of the back-up anesthetic nurse during the procedures proportion of surgical procedures requiring at least one intervention of the nurse
patient pre-surgical stress | baseline
  auto-assessment of stress level using a 0 to 10 (maximum stress) scale
pain during surgical procedure | within 10 minutes after surgery
  retrospective auto-assessment of patient pain using a 0 to 10 (maximum pain) scale
patient satisfaction | within 10 minutes after surgery
  auto-assessment of patient satisfaction using a 0 to 10 (fully satisfied) scale
incidence rate of each of the events included in the primary outcome | during surgical procedure
  incidence rate of blood pressure > 200 mmHg on 2 consecutive measures (automatic measure every 3 minutes) incidence rate of cardiac frequency < 45/min for at least 1 mn incidence rate of SaO2 <85% for at least 1 mn incidence rate of poor operating conditions (rated < 7 by the surgeon, on a numeric scale from 0 to 10 (excellent conditions)
patient agitation | within 10 minutes after surgery
  assessed by the surgeon using a 0 to 10 (very agitated) scale
operating conditions | within 10 minutes after surgery
  auto-assessment by the surgeon of the operating conditions, on a 0 to 10 (excellent conditions) scale and on a 0 to 10 (completely safe) scale
working conditions | at the end of a working day
  auto-assessment of working conditions by the anesthetic nurses, on a 0 to 10 (excellent) scale and on a 0 to 10 (completely safe) scale

OTHER OUTCOMES:
revision surgery | 24 hours after baseline
  incidence rate of revision surgery within 24 hours
efficiency of the centralised monitoring of anesthesic surveillance | during surgical procedure
  assessment of costs
patient baseline pain | baseline
  auto-assessment of patient pain before surgery on a 0 to 10 (maximum pain) scale

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Michel DEVYS, MD, Principal Investigator — Fondation Ophtalmologique Adolphe de Rothschild
Locations (1):
- Fondation Ophtalmologique Adolphe de Rothschild, Paris, Île-de-France Region, France

REFERENCES:
- [Result] Clariot S, Moures JM, Lopes L, Gatinel D, Gabison E, Nicolaos G, Salomon L, Devys JM. Centralized monitored anesthesia care by nurse anesthetist for cataract and glaucoma surgery in a 1:3 ratio: a non-inferiority study. Minerva Anestesiol. 2025 Mar;91(3):176-183. doi: 10.23736/S0375-9393.24.18455-6. Epub 2024 Dec 4. PMID 39630143